CLINICAL TRIAL: NCT07026851
Title: Pilot Study to Establish a Repertoire of Megakaryocyte Markers, Quantifiable by Spectral Flow Cytometry, in Bone Marrow and Circulating in Patients Undergoing Cardiac Surgery for Bypass Grafting
Acronym: EPIMéCA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0106; ID-RCB : 2025-A00744-45 (Other: Agence National de Sécurité du Médicament)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Surgery for Bypass Grafting
Keywords: Megakaryocytes; flow cytometry; cardiac surgery
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and bone marrow sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Bypass Grafting Patients Undergoing Bone Marrow and Blood Megakaryocyte Phenotyping
  Interventions: Biological: Blood and bone marrow sampling

INTERVENTIONS:
Biological: Blood and bone marrow sampling — This intervention involves the collection of peripheral blood before and 3 days after coronary artery bypass grafting (CABG), as well as a one-time collection of bone marrow sample during sternotomy.
  Samples are analyzed using spectral flow cytometry to characterize the phenotype and maturation stages of circulating and medullary megakaryocytes using a panel of specific surface antibodies.

SUMMARY:
Megakaryopoiesis, the mechanism of blood platelet production, is difficult to assess in clinical practice as it relies solely on microscopic description. Recent studies described the presence of emergency megakaryopoiesis bypassing the classical maturation stages under certain conditions. Circulating megakaryocytes were identified in inflammatory and hemostatic conditions. The aim of this study is to characterize the phenotype of medullar and circulating megakaryocytes by flow cytometry during and after coronary artery bypass grafting.

DETAILED DESCRIPTION:
Blood platelets, known for their role in primary hemostasis, are produced through the fragmentation of bone marrow megakaryocytes (MKs). In recent years, the characterization of new platelet functions, particularly in innate immunity and inflammatory processes, has reshaped the paradigm of sequential bone marrow megakaryopoiesis. Indeed, numerous studies provide evidence of a more direct, so-called "emergency" platelet production, which bypasses the successive stages of megakaryocyte differentiation. Furthermore, megakaryopoiesis may not be exclusively marrow-based; splenic and pulmonary sites are also described, along with circulating megakaryocytes in peripheral blood. These circulating megakaryocytes are gaining interest due to their easier accessibility and specific characteristics, notably pro-inflammatory properties.

However, to date, clinical practice analysis of megakaryocytes remains limited to simple microscopic description. Given recent observations as outlined above, a more precise and in-depth description of megakaryocytes, whether marrow-based or blood-based, appears essential for understanding pathophysiological mechanisms. Flow cytometry (FC) coupled with spectral technology overcomes the traditional limitations of FC. This technique has allowed our team to describe different stages of marrow megakaryocyte maturation using a murine model of platelet pathology.

In this context, cardiac surgery with extracorporeal circulation for coronary artery bypass grafting could serve as a model for inflammatory and hemostatic challenges. Post-procedural thrombocytopenia is common and is partly correlated with the duration of extracorporeal circulation (ECC), which could be associated with thrombo-inflammation responsible for acute kidney injury or stroke. Due to both the physiological bone marrow challenge posed by this procedure and the ease of bone marrow collection inherent to this technique, this situation seems well-suited for conducting this feasibility study.

Currently, no study has described the impact of megakaryocyte phenotype on platelet changes induced by cardiac surgery, whether these changes are purely quantitative or associated with a deleterious pro-inflammatory post-procedural context.

Based on these elements, combined with the expertise we have gained from studying the megakaryocyte/platelet axis in small animals using spectral flow cytometry, we propose:

* To validate the established antibody panel that allows the identification and quantification of the different maturation stages of bone marrow megakaryocytes,
* To apply this panel to circulating megakaryocytes before and after the surgical procedure,
* To correlate the observations with the potential inflammatory signature for each patient.

The rationale for this pilot study is to consider circulating megakaryocytes as a new, accessible, and highly specific indicator of thrombo-inflammatory processes.

ELIGIBILITY:
Inclusion Criteria:

- Age over 18

* Indication for programmed cardiac surgery, specifically coronary artery bypass grafting with sternotomy
* Up to date social security coverage
* Patients able to understand the purpose and constraints of the research project

Exclusion Criteria:

* Refusal to participate in the study,
* Pregnant and/or breastfeeding women (clinical interview),
* Unscheduled cardiac surgery, Acquired hematologic disorders (acute leukemia, lymphomas, myelodysplastic syndromes, and myeloproliferative syndromes)

  * Treatment with thrombopoietin receptor agonists
  * Treatment with anti-inflammatory (included corticoids) or/and immunosuppressors
  * Hematopoietic stem cell transplantation or organ transplantation
  * Active cancer with or without treatment (in remission, ongoing or treated within the last 6 months),
  * Palliative care patients
  * Any other type of cardiac surgery and previous sternotomy,
  * History of external thoracic radiotherapy,
  * Patient under legal protection (curatorship, guardianship or safeguard of justice)
  * Patients with ongoing clinical trial requiring collection of additional blood or bone marrow samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Department of Cardiovascular Surgery at Rangueil Hospital, Toulouse University Hospital (CHU Toulouse), during scheduled hospitalizations for elective coronary artery bypass grafting. The study population consists of adult patients programmed for cardiac surgery, specifically coronary artery bypass grafting with sternotomy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Phenotype of bone marrow and circulating megakaryocytes | Day of surgery
  Circulating and bone marrow megakaryocytes will be analyzed using spectral flow cytometry on samples collected during coronary artery bypass surgery. Cells will be labeled with a panel of specific surface antibodies . Megakaryocytes will be classified by maturation stage (multipotent progenitor [MPP], common myeloid progenitor [CMP], megakaryocyte-erythrocyte progenitor [MEP], pro-megakaryocyte [proMK], immature megakaryocyte [imMK], mature megakaryocyte [MK]) and specialization status (specialized MKs).

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Ribes, Principal Investigator — Toulouse, Rangueil Hospital
Locations (1):
- Toulouse University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No